CLINICAL TRIAL: NCT03358888
Title: Prolonged Multimodal Analgesia for Post-Discharge Pain Control After Primary Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017- Chen
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Active Comparator)
  Interventions: Drug: Standard of Care
- Multi-modal with as needed opioids (Active Comparator)
  Interventions: Drug: Multi-modal with as needed opioids
- Multi-modal with one week of opioids offered (Active Comparator)
  Interventions: Drug: Multi-modal with one week of opioids offered

INTERVENTIONS:
Drug: Multi-modal with as needed opioids — Multi-modal with as needed oxycodone and tramadol provided for break-through pain
  Arms: Multi-modal with as needed opioids
Drug: Multi-modal with one week of opioids offered — Multi-modal with only one week of oxycodone and tramadol provided for emergency pain relief only
  Arms: Multi-modal with one week of opioids offered
Drug: Standard of Care — This arm follows standard of care post-operative pain management with oxycodone, tramadol, and acetametophin
  Arms: Standard of Care

SUMMARY:
This is a prospective, three-arm, comparative study with a provider-crossover design. The first arm will comprise the standard of care pain regimen after discharge, which comprises PRN oxycodone, tramadol, and acetaminophen. The second arm will comprise a multimodal pain regimen; however, patients will still be routinely provided PRN oxycodone and tramadol to use on an as needed basis. The third arm will comprise a multimodal pain management protocol, which does not routinely allow for opioid consumption. However, patients will be provided a one week supply of oxycodone and tramadol for emergency pain relief only.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral, primary cementless THA with underlying diagnosis of osteoarthritis.
* ASA I - III
* Spinal anesthesia
* Male and Female over 18 who are willing and able to provide informed consent

Exclusion Criteria:

* Opioid use within 3 months prior to surgery
* General anesthesia
* Non-english speaking
* ASA IV or greater
* Allergy/contraindications to protocol medications
* Renal insufficiency with Cr > 2.0 or hepatic failure
* Sensory/motor disorder involving the operative limb
* Planned or unplanned discharge to rehab
* Length of stay >3 days
* Revision or conversion THA
* Cigarette smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
total opioid consumption | total consumption calcuated from surgery date through 30 days post-op
Pain | 30 days post-operative
  Pain as reported by Visual Analog Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Fleischman AN, Tarabichi M, Foltz C, Makar G, Hozack WJ, Austin MS, Chen AF; Opioid Prescription in Orthopedic Surgery after Discharge Research Group. Cluster-Randomized Trial of Opiate-Sparing Analgesia after Discharge from Elective Hip Surgery. J Am Coll Surg. 2019 Oct;229(4):335-345.e5. doi: 10.1016/j.jamcollsurg.2019.05.026. Epub 2019 Jun 5. PMID 31176028